CLINICAL TRIAL: NCT01815970
Title: Does Pulmonary Rehabilitation Reduce Neuromechanical Uncoupling of the Respiratory System in COPD
Brief Title: Does Pulmonary Rehabilitation Improve Breathing of COPD Patients
Acronym: PR-COPD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study never initiated.
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jordan Guenette, Assistant Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H13-00591
Record Dates: First submitted 2013-03-11; First posted 2013-03-21 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: dyspnea; exercise; neuromechanical uncoupling; COPD; pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulmonary Rehabilitation (Experimental): 8 weeks of Pulmonary Rehabilitation
  Interventions: Behavioral: Pulmonary Rehabilitation

INTERVENTIONS:
Behavioral: Pulmonary Rehabilitation — 8 weeks of Pulmonary Rehabilitation including exercise and COPD related education.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is the fourth leading cause of death world-wide. Dyspnea (i.e., sensations of breathlessness) is the hallmark symptom of patients with this disease. Pulmonary rehabilitation programs that incorporate exercise training remain the most effective non-pharmacological method of reducing dyspnea in COPD, however it is not understood how exercise training relieves dyspnea. Accordingly, the purpose of this study is to determine if pulmonary rehabilitation can reduce the disparity between the drive to breathe and the breathing response in patients with COPD and to determine if this reduction is associated with improvements in dyspnea during exercise.

The investigators hypothesise pulmonary rehabilitation will reduce dyspnea at a standardized work rate and this reduction will be directly related to an improvement in the breathing response.

DETAILED DESCRIPTION:
The purpose of this study is to determine if 8 weeks of pulmonary rehabilitation can reduce neuromechanical uncoupling (a disparity between the effort/drive to breathe and the breathing response) in patients with COPD and to determine if this reduction is associated with improvements in both the intensity and qualitative dimensions of dyspnea during exercise.

Pulmonary rehabilitation is an exercise and education intervention designed to help patients cope with their dyspnea, and exercise effectively. Pulmonary rehabilitation programs that incorporate exercise training are the most effective non-pharmacological method of reducing dyspnea in COPD. However, the precise mechanisms of dyspnea relief following exercise training are still unknown. Understanding the pathophysiologcal underpinnings of this debilitating symptom is critical in order to develop effective symptom-based strategies for dyspnea management.

Participants with COPD will report to the exercise laboratory on 3 separate visits. Visit 1 will serve as an initial screening visit whereby participants will provide written informed consent prior to familiarization of all testing procedures and symptom scales followed by completion of an incremental cycle exercise test. The remaining 2 experimental visits will be conducted immediately before and after 8 weeks of pulmonary rehabilitation. Visits 2 and 3 will include: symptom-related questionnaires, pulmonary function tests, functional ability test and a constant-work rate (CWR) cycle exercise test at 75% of the maximal work rate achieved during visit 1. The CWR cycle exercise tests will be performed with the instrumentation of an esophageal catheter and detailed physiological and sensory measurements will be obtained on both visits. The comparison of data from visits 2 and 3 will address the investigators' hypotheses.

Study Participants: The study will include 12 COPD participants in total. Pulmonary Rehabilitation: The pulmonary rehabilitation program provides education and exercise training for patients with chronic lung disease to assist them with symptom management and improve their daily ability to function. The 8 week program involves 3 visits per week for 2 hours each visit (1 hour education and 1 hour exercise training). The pulmonary rehabilitation program is usual care for all participants in this study.

Exercise Protocol: A symptom-limited incremental exercise test will be performed on visit 1 using an electronically braked cycle ergometer according to recommended guidelines. The test will consist of steady-state rest for 10 minutes, a 1 minute warm-up at 0 watts, and 10 watt stepwise increases in work rate every minute until symptom-limitation. The CWR test performed on visits 2 and 3 will consist of a 1 minute warm-up followed by an increase in work rate to 75% of the maximum incremental work rate.

Measurements Pulmonary Function: Spirometry, plethysmography, diffusing capacity, and maximum respiratory pressures will be performed on visit 1 according to standard recommendation. Visits 2 and 3 will include spirometry, plethysmography, and maximum respiratory pressures. A commercially available cardiopulmonary testing system (Vmax 229d with Autobox 6,200 DL; SensorMedics, Yorba Linda, CA) will be used, and all measurements will be expressed as percent of predicted normal values.

Dyspnea Evaluation: Dyspnea intensity (defined as "the sensation of laboured or difficult breathing") and perceived leg discomfort will be evaluated at rest, every minute during exercise, and at peak exercise using the modified 10-point Borg scale on all testing visits. Participants will be asked to describe their dyspnea during exercise prior to the intensity ratings and at end-exercise using the following 3 descriptors: (1) "my breathing requires more work and effort" (work and effort); (2) "I cannot get enough air in" (unsatisfied inspiration); (3) "I cannot get enough air out" (unsatisfied expiration). None to all 3 of the descriptors can be chosen at any one time. Upon exercise cessation, participants will be asked to verbalize their main reason(s) for stopping exercise (i.e., breathing discomfort, leg discomfort, combination of breathing and legs, or some other reason) and to select qualitative descriptors of breathlessness using an established questionnaire. Pre- to post-intervention changes in dyspnea will also be assessed with the Transition Dyspnea Index.

Cardio-respiratory Responses to Exercise: Standard cardio-respiratory measures will be recorded on a breath-by-breath basis and averaged over 30-second epochs, including minute ventilation (V'E), oxygen consumption (VO2), carbon dioxide production (CO2), partial pressure of end-tidal CO2, (tidal volume) VT, and breathing frequency (Vmax 229d with Autobox 6,200 DL; SensorMedics, Yorba Linda, CA). Operating volumes (i.e., end-expiratory and end-inspiratory lung volumes) will be derived from dynamic inspiratory capacity (IC) manoeuvres as previously described 26. For safety purposes, electrocardiography will be monitored using a 12-lead electrocardiogram (ECG), blood pressure will be measured using a manual sphygmomanometer, and arterial oxygen saturation will be monitored using pulse oximetry. Exercise tests will be terminated based on established criteria as per American College of Sports Medicine guidelines.

Respiratory Mechanics: Diaphragmatic electromyography (EMGdi) will be measured using a multi-pair electrode catheter that combines two balloons for measuring esophageal and gastric pressures. Lidocaine spray or gel (a local anaesthetic) will be used to freeze the participant's nose and back of their throat. After which, while the participant sips water through a straw, an experienced technician will insert the catheter through the participants nose and into their stomach via their esophagus. The catheter will be positioned based on the strength of EMGdi signal during spontaneous breathing. The raw EMGdi signal will be converted to a root mean square (RMS). The maximum RMS for each inspiration will be determined between QRS complexes to avoid the influence of ECG artefact 30. Maximal EMGdi (EMGdimax) will be obtained during IC, sniff and maximal inspiratory pressure manoeuvres. The ratio of EMGdi to EMGdimax will be used as an index of neural respiratory drive. The ratio between VT and vital capacity (VC) will be used to represent the mechanical response of the respiratory system. Normalizing for EMGdimax and VC allows the stimulus intensity to be standardized and compared across individuals. Thus neuromechanical uncoupling of the respiratory system will be determined as the ratio (or interaction) between neural drive and the mechanical response of the respiratory system (EMGdi/EMGdimax : VT/VC).

The mechanical work of breathing (WOB) will be determined using modified Campbell diagrams as used previously. Chest wall compliance will be obtained from the literature and positioned as previously described. The WOB will be partitioned into its resistive and elastic components. This data will be compared to the WOB data in previous COPD studies.

Muscle oxygenation and hemodynamics: Muscle oxygenation will be noninvasively monitored using near infrared spectroscopy. A four-channel continuous-wave near-infrared spectroscope (Oxymon M III, Artinis Medical Systems, BV, The Netherlands) will be used to determine oxyhemoglobin, deoxyhemoglobin, and total hemoglobin by measuring light attenuation at 760 and 864 nm wavelengths, and analyzed using algorithms based on the modified Beer-Lambert law. This data will be used for descriptive exploratory purposes as limited data exists on the muscle oxygenation of the legs (vastus lateralis) and respiratory muscles (sternocleidomastoid, parasternal, and intercostals) in COPD patients.

Inflection Point of the VT and V'E Relationship: VT data will be averaged over 30-second epochs and will be plotted against V'E at rest and throughout all exercise intensities for each individual participant. The point at which VT deviates from linearity and begins to plateau will be defined as the inflection point of the VT and V'E relationship. Two different observers will determine the inflection point for each participant during the incremental exercise test by examining individual Hey plots.

Statistical Analysis: Data will be presented as means ± SD unless otherwise specified. Pre and post-pulmonary rehabilitation descriptive characteristics, exercise responses, and Borg ratings at standardized evaluation points (10 watt increments, VT/V'E inflection, and peak) will be compared using paired t-tests with Bonferroni corrections where appropriate. Pearson correlation coefficients will be used to examine the association between measured variables: neuromechanical uncoupling, breathing pattern, operational lung volumes, Borg ratings, and exercise variables. Reasons for stopping exercise and qualitative descriptors of dyspnea will be analyzed as frequency statistics and compared between pre and post pulmonary rehabilitation using the McNemar's exact test at standardized 10 watt increments in work-rate, VT/V'E inflection, and peak exercise. A P-value less than 0.05 will be regarded as statistically significant. Statistical analysis of the data will be performed using Stata v11.2 (StataCorp, Texas, USA).

ELIGIBILITY:
Inclusion Criteria:

* A physician diagnosis of moderate-to-severe COPD
* Stable clinical COPD status (no history of an acute exacerbation requiring antibiotics or prednisone in the past 4 weeks)
* Post-bronchodilator Forced Expiratory Volume in 1 second (FEV1.0) ≥ 30 - < 80% predicted and FEV1.0/Forced Vital Capacity ratio < 0.7
* Body mass index > 18 or < 35 kg/m2
* Able to read and understand English

Exclusion Criteria:

* Concurrent participation in or recent completion (<6 weeks) of pulmonary rehabilitation
* An ulcer or tumor in their esophagus, or a nasal septum deviation (as reported by the participant)
* Had recent nasopharyngeal surgery
* Have a cardiac pacemaker
* Allergies to latex and sensitivities to local anesthetics
* Uncontrolled hypertension
* Diagnosis of diabetes
* Previous physician diagnosis of cardiovascular disease including: angina, acute coronary syndrome, heart failure, cerebrovascular disease, thromboembolic disease, peripheral vascular disease
* Other chronic lung disease including: asthma, interstitial lung disease, or pulmonary hypertension
* Chronic hepatic disease, chronic renal disease, or other systemic inflammatory disease
* Use of chronic oral steroids
* Dementia or uncontrolled psychiatric illness
* A disease other than COPD that could contribute to dyspnea or exercise limitation
* Contraindications to clinical exercise testing

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in neuromechanical uncoupling | Parameters will be measured during the 3 visits, at rest and during exercise. Visits 1 & 2 will be 48 hrs apart and within 2 weeks prior to the 8 week pulmonary rehabilitation (PR). Visit 3 will occur within 2 weeks after the completion of the PR.
  The relationship between the neural drive (or effort) to breathe and the corresponding mechanical response of the respiratory system.

SECONDARY OUTCOMES:
Dyspnea | Parameters will be measured during the 3 visits, at rest and during exercise. Visits 1 & 2 will be 48 hrs apart and within 2 weeks prior to the 8 week pulmonary rehabilitation (PR). Visit 3 will occur within 2 weeks after the completion of the PR.
  Intensity (BORG scale) and qualitative dimensions (dyspnea descriptors) of dyspnea.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan A Guenette, Ph.D., Principal Investigator — UBC James Hogg Research Centre/ UBC Dept. Physical Therapy
Locations (1):
- UBC James Hogg Research Centre, St. Paul's Hospital, Vancouver, British Columbia, Canada